CLINICAL TRIAL: NCT05538468
Title: Investigation of the Relationship Between Depression, Postural Control, Pain, Affected Side and Kinesiophobia in Stroke Patients
Brief Title: Kinesiophobia in Stroke Patients and Affecting Factors
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate Professor Doctor, Inonu University
Other Study IDs: 2019/3-22
Record Dates: First submitted 2022-01-13; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-01

CONDITIONS: Kinesiophobia; Stroke Patients
Keywords: Kinesiophobia; stroke patients; Pain; Postural control; Depression
MeSH Terms: conditions — Kinesiophobia; Pain; Depression | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke Patients Group: The kinesiophobia scores of the patients were evaluated by (Tampa Kinesiophobia Scale) and (Visual Analog Scale- Kinesiophobia Assessment), depression severity (Beck Depression Inventory), postural control (Postural Assessment Scale), pain severity (Visual Analog Scale).
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Thirty stroke patients were included in the study. After the demographic information was obtained from all patients who accepted to participate in the study by complying with the inclusion criteria; The kinesiophobia scores of the patients were evaluated, depression severity, postural control and pain severity.

SUMMARY:
It was aimed to determine the presence of kinesiophobia that will affect the treatment in stroke patients and to investigate the relationship between these factors and kinesiophobia by examining factors such as postural control, depression, pain, and affected side that may cause kinesiophobia.

DETAILED DESCRIPTION:
Objective: This study was planned to investigate the relationship between depression, postural control, pain, affected side and kinesiophobia in stroke patients. Material and Method: Thirty patients aged between 25-70 years who had a stroke at the earliest 6 months and who Functional Ambulation Scale were level 2 and above according to the were included in the study. Patients were selected by random sampling method from the relevant population. Demographic data were obtained from all subjects who met the inclusion criteria. Patients were evaluated Kinesiophobia scores (Tampa Kinesiophobia Scale (TKÖ) and VAS-Kinesiophobia Assessment), depression severity (Beck Depression Inventory), postural control loss (PASS) and pain severity (VAS).

ELIGIBILITY:
Inclusion Criteria:

* individuals who were diagnosed with hemiplegia or hemiparesis after SVO,
* at least 6 months after SVO,
* who were Level 2 and above according to the Functional Ambulation Classification,
* who wanted to participate in the study voluntarily

Exclusion Criteria:

* Anyone with a major neurological or rheumatological pathology (polyneuropathy, parkinson's, multiple sclerosis, rheumatoid arthritis, etc.)
* Affecting the musculoskeletal system other than stroke
* Who does not allow mental evaluation, cannot fill in the scales,
* is illiterate, has aphasia, has a history of falling,
* have any cardiac problems,
* amputation in the lower extremities,
* those with active malignancy and related chemo/radiotherapy,
* the presence of accompanying lower motor neuron or peripheral nerve lesion,
* any musculoskeletal problem and related pain (lumbar disc herniation, meniscus, etc.),
* ındividuals with shoulder subluxation, shoulder-hand syndrome
* those who refused to participate in the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients who were level 2 and above according to the Functional Ambulation Classification were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia Assessment | 6 mounts
  VAS Kinesiophobia Assessment were used. The Visual Analog Scale was used as the second method in the assessment of kinesiophobia. A scale is drawn on a 10-centimeter (cm) horizontal line to show the start as 0 (no fear of movement) and the end as 100 (violent fear of movement). They were asked to stand up just before starting the exercise and to mark the severity of the fear of movement they felt at that moment on the scale.
Kinesiophobia Assessment | 6 mounts
  Tampa Kinesiophobia Scale were used. The Tampa Kinesiophobia Scale (TKS) is one of them, and it's commonly used in the literature to assess kinesiophobia. It has 17 questions designed to assess fear of moving.
Pain Assessment | 6 mounts
  Pain Assessment Visual Analogue Scale (VAS) was used. On a 10-centimeter (cm) horizontal line, start 0 (no pain) and finish 10 (unbearable pain) are marked and the subjects were asked to place a mark on this horizontal line according to the degree of pain they felt. The point marked on the line was then measured with the help of a ruler and recorded as the VAS value in cm.
Postural Control Assessment | 6 mounts
  Postural Assessment Scale for Stroke Patients (PASS) was used. The scale, which consists of 12 items, is grouped at 4 different levels (0-3). It is a 2-part scale that assesses the ability to maintain the posture (5 items) and change it (7 items).
Depression Severity Assessment | 6 mounts
  Depression Severity Assessment, The Beck Depression Inventory (BDI) was employed, which consists of 21 questions. The scale has a range of 0 to 84 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No